CLINICAL TRIAL: NCT06617442
Title: Esophageal Safety of High and Very High Power Short Duration Pulmonary Vein Isolation: a Randomized Comparison of the 50W and 90W Power Settings
Acronym: HPSD-Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Nandor Szegedi, Assistant Professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8088-2/2022/EÜIG
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF); Esophageal Perforation; Esophageal Perforation, Traumatic
Keywords: Pulmonary Vein Isolation; PVI; HPSD; High Power Short Duration; Esophageal injury
MeSH Terms: conditions — Atrial Fibrillation; Esophageal Perforation

STUDY DESIGN:
Intervention Model Description: Randomized, open label
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 90W (Experimental): Pulmonary vein isolation performed using very-high power short duration applications (90-watt applications lasting 4 seconds).
  Interventions: Procedure: Pulmonary vein isolation
- 50W (Active Comparator): Pulmonary vein isolation performed using high power short duration applications (50-watt applications guided by ablation index).
  Interventions: Procedure: Pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation — First pulmonary vein isolation performed for atrial fibrillation.

SUMMARY:
Pulmonary vein isolation (PVI) is the most effective means of maintaining sinus rhythm in atrial fibrillation (AF), while a widely used approach to PVI is point-by-point radiofrequency (RF) catheter ablation. High power short duration (HPSD) and very high power short duration e.g., 90W and 4 sec) are increasingly popular technologies, featuring higher power and shorter application durations compared to previous methods. vHPSD offers similar efficacy to HPSD, while further reducing procedure times. Atrioesophageal fistula (AEF) is a rare but deadly complication of PVI, while endoscopically detected esophageal lesions are surrogate markers for the risk of AEF. Furthermore, thermal complications include vagal lesions leading to gastroparesis. While there is considerable data on the thermal safety of HPSD technology, most studies of vHPSD focus on efficacy and a direct comparison in terms of esophageal safety is lacking. In this randomized, single-center study, we aim to compare the thermal safety of vHPSD to HPSD. Furthermore, we aimed to determine the anatomical and biophysical factors that predict thermal injury. Patients undergoing their first PVI for AF are randomized to either HPSD or vHPSD power setting. The primary endpoint of the study is the composite of esophageal mucosal lesion and gastroparesis, as assessed at the post-procedural endoscopy within 15 days after the PVI.

ELIGIBILITY:
Inclusion Criteria:

- Patients with paroxysmal or persistent atrial fibrillation undergoing their first pulmonary vein isolation procedure

Exclusion Criteria:

* Additional ablation performed outside PVI
* Contraindications to postoperative upper endoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Thermal injury detected during post-procedural endoscopy | Post-procedural endoscopy was performed within 15 days after the procedure.
  Composite of esophageal ulcer or erosion and gastric hypomotility.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University Heart and Vascular Center, Budapest, Hungary, Hungary

IPD SHARING:
Plan to Share IPD: No